CLINICAL TRIAL: NCT06582446
Title: Whole-pelvis Hypofractionated Radiotherapy Combined With Dose-escalation to the Prostate and Androgen Deprivation Therapy in Primary Localized, NCCN and MMAI High-risk Prostate Cancer - a Prospective, Single-arm, Phase II Study
Brief Title: Artificial Intelligence to Personalize Prostate Cancer Treatment (the HypoElect Trial)
Acronym: HypoElect
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: German Oncology Center, Cyprus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-PRC-015; U1111-1310-7485 (Other: World Health Organization Universal Trial Number (UTN))
Record Dates: First submitted 2024-07-31; First posted 2024-09-03 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; multimodal AI; radiotherapy; phase II
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Androgen Antagonists; Goserelin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single experimental arm (Experimental): RT prostate (HDR brachytherapy): 15 Gy (D90) in 1 fraction HDR RT prostate
  EBRT elective pelvis (Ultra-hypofractionated RT - UHF): 25 Gy in 5 Gy per fraction
  Technique: IMRT/IGRT/HDR brachytherapy
  Duration: 6 fractions, 3 weeks
  Androgen deprivation therapy (ADT) - Goserelin: all patients receive ADT; luteinising-hormone-releasing hormone agonists or antagonists for 24 months
  Follow-up (FU) per patient: minimum FU time is 5 years (60 months), the study ends when the last enrolled patients reaches 60 months of FU time
  Further FU: by the end of this clinical trial it will be decided whether further FU is necessary, amendment to this clinical trial protocol will be done in appropriate time
  Interventions: Drug: Androgen Deprivation Therapy (ADT) - Goserelin; Radiation: High-Dose-Rate Interstitial Brachytherapy (HDR BRT); Radiation: radiotherapy

INTERVENTIONS:
Drug: Androgen Deprivation Therapy (ADT) - Goserelin — The patients under ADT and the patients who will receive the ADT during the study will be included in the trial.
  * ADT will be applied for 24 months in total
  * ADT must be given concurrently and adjuvant
Radiation: High-Dose-Rate Interstitial Brachytherapy (HDR BRT) — HDR BRT Procedure will be performed using transperineal catheter implantation under transrectal US-guidance performed under anesthesia, spinal or general with patient in high lithotomy position.)
Radiation: radiotherapy — EBRT prostate + elective pelvis (Ultra-hypofractionated): 25 Gy in 5 Gy per fraction

SUMMARY:
A prospective, single-arm phase II study is the individualization of RT for patients with high-risk localized PCa based on multimodal artificial intelligence (MMAI). All patients will receive the current standard of care: (i) a dose escalation to the prostate via HDR brachytherapy, (ii) two years of ADT and (iii) whole-pelvis UHF-RT (5 fractions).

DETAILED DESCRIPTION:
Prostate cancer (PCa) is the most frequent diagnosed malignancy in male patients in Europe and radiation therapy (RT) is a main treatment option. For primary high-risk localized PCa patients, NCCNv4.2023 guidelines recommend normo- or hypofractionated RT to the prostate ± the elective pelvic lymphatics and systemic treatment in terms of ADT. Although the standard of care, the benefit of this therapy regimen is controversially discussed: the benefit of (i) an RT dose escalation using brachytherapy (2) or focal dose escalated RT(3) or (ii) an elective RT of the pelvic lymph nodes (1) is not finally proven yet. In parallel, first studies proposed a reduction in treatment fractions in terms of ultra-hypofractionated RT (UHF-RT) (4).

The aim of this prospective, single-arm phase II study is the individualization of RT for patients with high-risk localized PCa based on MMAI. All patients will receive the current standard of care: (i) a dose escalation to the prostate via HDR brachytherapy, (ii) two years of ADT and (iii) whole-pelvis UHF-RT (5 fractions).

For the HypoElect patients we expect no significant differences in toxicity rates compared to the randomized controlled POP-RT trial (1) which treated the patients with moderately-hypofractionated RT to the prostate and the elective pelvic lymph nodes in parallel to 24 months of ADT. Secondary endpoints like relapse free survival, metastatic free survival, prostate cancer survival and overall survival will depict the oncologic efficacy in this patient cohort. Thus, the safety and oncologic outcome results of this study might be the first in this highly selected treatment group: NCCN high-risk, PSMA PET cN0/cM0 and MMAI high-risk. Considering the epidemiological importance of the PCa these results could have a significant socio-economic impact. In parallel a translational research program will address the identification of novel biomarkers to predict the treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate (histological confirmation can be based on tissue taken at any time, but a re-biopsy should be considered if the biopsy is more than 12 months old)
* Primary PCa (in PSMA-PET imaging and multiparametric magnetic resonance imaging (mpMRI)
* High- or very high-risk according to NCCNv1.2023 criteria
* Signed written informed consent for this study
* Age >18 years
* Previously conducted PSMA-PET/CT, mpMRI or PSMA-PET/MR
* MMAI high-risk
* ECOG Performance score 0 or 1
* IPSS Score ≤15

Exclusion Criteria:

* Prior radiotherapy to the prostate or pelvis
* Prior radical prostatectomy
* Prior focal therapy approaches to the prostate
* Evidence of pelvic nodal disease (cN+) in mpMRI and/or PSMA-PET/CT
* Evidence of distant metastatic disease (cM+) in mpMRI and/or PSMA-PET/CT
* Time gap between the beginning of any systemic therapyADT and conduction of PSMA-PET scans is >2 months
* Evidence of cT4 disease in mpMRI and/or PSMA-PET/CT
* PSA >50 ng/ml prior to starting of systemic therapy
* Expected patient survival <5 years
* Bilateral hip prostheses or any other implants/hardware that would introduce substantial CT artifacts
* Contraindication to undergo a MRI scan
* Contraindication to undergo HDR brachytherapy (brachytherapy not feasible due to large prostate volume, prostate anatomy, tumor in distant seminal vesicles and/or unfit for anesthesia)
* Prostate surgery (TURP or HOLEP) with a significant tissue cavity or prostate surgery (TURP or HOLEP) within the last 6 months prior to randomization
* Medical conditions likely to make radiotherapy inadvisable e.g. acute inflammatory bowel disease, hemiplegia or paraplegia
* Previous malignancy within the last 2 years (except basal cell carcinoma or squamous cell carcinoma of the skin), or if previous malignancy is expected to significantly compromise 5 year survival
* Any other contraindication to external beam radiotherapy (EBRT) to the pelvis
* Participation in any other interventional clinical trial within the last 30 days before the start of this trial
* Simultaneous participation in other interventional trials which could interfere with this trial; simultaneous participation in registry and diagnostic trials is allowed
* Patient without legal capacity who is unable to understand the nature, significance and consequences of the trial
* Known or persistent abuse of medication, drugs or alcohol

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males with prostate cancer. Eligibility is based on histologically confirmed adenocarcinoma of the prostate
Enrollment: 30 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
cumulative GU toxicity | two years
  Primary endpoint is cumulative GU toxicity according to RTOG grading after minimum FU time of two years.

SECONDARY OUTCOMES:
Time to local or regional failure | two and five years after RT
  Time to local or regional failure; after end of RT. Local or regional recurrences have to be confirmed by PSMA-PET or mpMR imaging. For the diagnosis of local failure a verification via biopsy is warranted.
MMAI classifier | 5-year and 10-year risk prediction of distant metastasis and 10-year risk of prostate-specific mortality.
  Prognostic influence of MMAI classifier for outcome; the ArteraAI Prostate Test score (ranging from 0.0 to 1.0)
Testosterone | assessment at 6,9,12,18 and 24 months after randomization (± 14 days for each visit) and at 30, 36, 42, 48, 54, 60 months after Ultra-hypofractionated RT - UHF (± 1 month
  Testosterone recovery is to be done through blood test
Metastatic free survival (MFS) | two and five years after RT
  MFS after end of RT, (all metastases have to be confirmed by PSMA-PET/CT or mpMR imaging)
Overall Survival (OS) | 1, 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54 and 60 months after RT
  OS after end of RT
Prostate cancer specific survival (PCSS) | 1, 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54 and 60 months after RT
  PCSS after end of RT
Biochemical failure | two and five years after RT
  Time to biochemical failure after end of RT (phoenix definition)
Quality of Life (QoL) | Assessments at 6, 9,12, 18, and 24 months after randomization (± 14 days for each visit) and at 30, 36, 42, 48, 54, 60 months after Ultra-hypofractionated RT - UHF (± 1 month)
  Patient-reported outcome measures (PROMs) EPIC-26: the Expanded Prostate Cancer Index-Short form) with score: 0-100
QoL | Assessments at 6, 9,12, 18, and 24 months after randomization (± 14 days for each visit) and at 30, 36, 42, 48, 54, 60 months after Ultra-hypofractionated RT - UHF (± 1 month)
  Patient-reported outcome measures (PROMs) IIEF-5: The International Index of Erectile Function with score: 0-5
QoL | Assessments at 6, 9,12, 18, and 24 months after randomization (± 14 days for each visit) and at 30, 36, 42, 48, 54, 60 months after Ultra-hypofractionated RT - UHF (± 1 month)
  Patient-reported outcome measures (PROMs) IPSS: International prostate symptom score with score 0-5
Genitourinary (GU) acute toxicities | during, 1 and 3 months after RT
  Cumulative acute GU toxicities using the RTOG grading system (Radiation Therapy Oncology Group; with grade: 0-5, where 0 implies no toxicity and 5 implies a side effect related to death)
GU acute toxicities | during, 1 and 3 months after RT
  Cumulative acute GU toxicities using the CTCAE v5.0 criteria (the Common Terminology Criteria for Adverse Events criteria; with grade: 1-5 where 1 means asymptomatic or mild symptoms and 5 means death related to adverse event)
GU chronic toxicities | 6, 9, 12, 18 and 24 months after RT
  Cumulative chronic GU toxicities using the RTOG grading system (Radiation Therapy Oncology Group; with grade: 0-5, where 0 implies no toxicity and 5 implies a side effect related to death)
GU chronic toxicities | 6, 9, 12, 18 and 24 months after RT
  Cumulative chronic GU toxicities using the CTCAE v5.0 criteria (the Common Terminology Criteria for Adverse Events criteria; with grade: 1-5 where 1 means asymptomatic or mild symptoms and 5 means death related to adverse event)
Gastrointestinal (GI) acute toxicities | during, 1 and 3 months after RT
  Cumulative acute GI toxicities using the RTOG grading system (Radiation Therapy Oncology Group; with grade: 0-5, where 0 implies no toxicity and 5 implies a side effect related to death)
GI acute toxicities | during, 1 and 3 months after RT
  Cumulative acute GU toxicities using the CTCAE v5.0 criteria (the Common Terminology Criteria for Adverse Events criteria; with grade: 1-5 where 1 means asymptomatic or mild symptoms and 5 means death related to adverse event)
GI chronic toxicities | 6, 9, 12, 18 and 24 months after RT
  Cumulative chronic GU toxicities using the RTOG grading system (Radiation Therapy Oncology Group; with grade: 0-5, where 0 implies no toxicity and 5 implies a side effect related to death)
GI chronic toxicities | 6, 9, 12, 18 and 24 months after RT
  Cumulative chronic GU toxicities using the CTCAE v5.0 criteria (the Common Terminology Criteria for Adverse Events criteria; with grade: 1-5 where 1 means asymptomatic or mild symptoms and 5 means death related to adverse event)
Dose contrainsts | during, 1 and 3 months after RT
  Feasibility to dose constraints for pelvic lymph nodes irradiation
  HDR-BT
  Prostate CTV=PTV Reference dose DR: 15 Gy (100 %) D90 ≥ 100 % V100 ≥ 95 % V150 ≤ 30 %
  Rectum (OAR) D2cc ≤ 75Gy EQD2(1.5) D1cc ≤ 70%
  Urethra (OAR) D0.1cc ≤ 115% D10 ≤ 110% D30 ≤ 105Gy EQD2(1.5)
Dose contrainsts | during, 1 and 3 months after RT
  Feasibility to dose constraints for pelvic lymph nodes irradiation
  Pelvic EBRT PTV, Constraint, Vol cc or % PTV P/SV, V95 ≥, 95 PTV LV, V95 ≥, 95 Dmax LV, max < 107 Dmax SIB, max < 107
  OAR: Rectum Constraint, Vol cc or % V18Gy < (%), 50 V20Gy < (%), 30 D1cc ≤ (Gy), 26
  OAR: Sigmoid Constraint, Vol cc or % V18Gy < (%), 50 V20Gy < (%), 30 D1cc ≤ (Gy), 26
  OAR: Bladder Constraint, Vol cc or % V18Gy < (%), 50 V20Gy < (%), 30 D1cc ≤ (Gy), 26
  OAR: Femoral Head L Constraint, Vol cc or % D10cc ≤ (Gy), 25
  OAR: Femoral Head R Constraint, Vol cc or % D10cc ≤ (Gy), 25
  OAR: Bowel Cavity (including sigmoid) Constraint, Vol cc or % V25Gy < (cc), 40 D1cc ≤ (Gy), 26
  OAR: Penile bulb Constraint, Vol cc or % Mean < (Gy), 20
Dose contrainsts | during, 1 and 3 months after RT
  Adherence to dose constraints for pelvic lymph nodes irradiation Interruptions of RT in days along with reasons
Dose contrainsts | during, 1 and 3 months after RT
  Adherence to dose constraints for pelvic lymph nodes irradiation Treatment not finished due to set-up problems (YES/NO) and reason

CONTACTS AND LOCATIONS:
Overall Officials: Iosif Strouthos, MD, Principal Investigator — German Medical Institute; Constantinos Zamboglou, MD, Principal Investigator — German Medical Institute
Locations (1):
- German Oncology Center, Limassol, Cyprus

IPD SHARING:
Plan to Share IPD: No